CLINICAL TRIAL: NCT06045858
Title: Safety and Efficacy of Apixaban Versus Warfarin in Peritoneal Dialysis Patients With Non Valvular Atrial Fibrillation: a Prospective, Randomised, Open-label, Blinded End-point Trial (APIDP2)
Acronym: APIDP2
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-164; 2023-507544-37-00 (EU CTIS Number)
Record Dates: First submitted 2023-09-04; First posted 2023-09-21 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Peritoneal Dialysis Complication
Keywords: peritoneal dialysis; atrial fibrillation; anticoagulation; randomized controlled trial
MeSH Terms: conditions — Atrial Fibrillation | interventions — Anticoagulants

STUDY DESIGN:
Intervention Model Description: a Haybittle sequential plan (PROC SEQDESIGN, SAS 9.4) with decision rule for better safety (larger than expected effect)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warfarin (Active Comparator): Warfarin (Coumadine): INR target [2.0-3.0]
  Interventions: Drug: Anticoagulation Agents
- Apixaban (Experimental): Apixaban (Eliquis) at 2.5mg, per os, twice a day
  Interventions: Drug: Anticoagulation Agents

INTERVENTIONS:
Drug: Anticoagulation Agents — anticoagulation in peritoneal dialysis patients with non valvular atrial fibrillation during one year

SUMMARY:
Introduction:

Several randomised controlled trials have demonstrated that novel oral anticoagulants (NOACs) are safer compared to vitamin K antagonists for the management of non valvular atrial fibrillation (NVAF) to prevent thromboembolic events, in the general population. There is a growing interest in the use of apixaban in patients with End-Stage Renal-Disease (ESRD) undergoing peritoneal dialysis but there is a lack of randomised data in this population.

Design: APIDP2 is a prospective parallel randomised, open-label, blinded endpoint trial.

Participants: Patients with ESRD undergoing chronic Peritoneal Dialysis who have NVAF.

Setting: A total of 178 participants will be recruited from 20 French peritoneal dialysis centers.

Intervention: Eligible patients will be randomly assigned to receive either apixaban at a reduced dose 2.5mg twice daily (dose determined with the previous pharmacokinetic study APIDP1 of apixaban in PD patients) or dose-adjusted to INR target [2-3] coumadin therapy. Anticoagulation to prevent thromboembolic events will be initiated or changed according to the randomisation for a duration of one year.

The primary outcome is a major or clinically relevant non-major bleeding from randomisation up to Month 12, assessed according to ISTH score. Secondary outcomes encompass an efficacy composite criterion combining stroke or TIA, cardiovascular death, and thrombosis including myocardial infarction cumulated at 12 months. Bleeding events will be also classified according to GUSTO and TIMI criteria and pharmacodynamics outcomes will evaluate the time within the INR target range of [2-3] in the warfarin arm over one year, and AntiXa apixaban activity in case of bleeding events and at 1, 6, and 12 months of follow-up in the apixaban arm.

Primary outcome analysis: To demonstrate that apixaban is safer than warfarin at one year, assuming two interim analyses after 60 and 118 patients, a bilateral alpha risk of 5% and a power of 80%, 178 patients are needed in this randomised trial (effect size found in the ARISTOTLE study among patients with CrCl [25-30]ml/min), i.e. 89 patients per group.

DETAILED DESCRIPTION:
The prevalence of AF in the general population is estimated to range around 1% depending on age, reaching 8% in patients over 80 years old. This prevalence is of 20% and 14% in patients on hemodialysis and peritoneal dialysis.

In addition, AF is associated with higher morbidity and mortality rates in patients with advanced chronic kidney disease, in contrast with patients with preserved kidney function, with a higher risk of both bleeding and clotting.

In the general population, the novel oral anticoagulants (NOACs) demonstrated a greater safety over warfarin and among 269 patients with CrCl (Creatinine Clearance) 25 to 30 mL/min included in ARISTOTLE trial: apixaban caused less bleeding than warfarin.

Furthermore, warfarin has been recognized as a risk factor for calcific uremic arteriolopathy (calciphylaxis), a rare yet serious complication. Additionally, patients in ESRD appear to have low adherence to warfarin therapy, with time of INR in target range of only 44 to 51% in three randomised controlled trials.

Considering the complex pathophysiology underlying the excess risk of stroke in patients with advanced CKD and the known complications of warfarin therapy, the use of NOACs in these populations may present an appealing alternative.

Four significant reviews conducted in 2022 and 2023, based on randomised controlled trials and cohort studies, assessed both thrombotic and bleeding outcomes associated with anticoagulant use in advanced chronic kidney disease. These reviews highlights the necessity for more randomised controlled trials (RCTs).

The two most significant cohorts to date that compared warfarin versus NOACs yielded important findings are:

* Siontis et al.: they conducted a study involving a larger cohort (2,351 versus 7,053) and found a reduction in major bleeding events with apixaban compared to warfarin, with similar efficacy in dialysis patients.
* Wetmore et al.: they included 3,130 patients versus 9,086, and also found a reduction in major bleeding events with apixaban compared to warfarin in dialysis patients, while maintaining similar efficacy.

In 2023, a thirth cohort study was published, involving 4,313 apixaban users with stage 4 and 5 kidney disease. This study found that the use of 5mg apixaban was associated with a higher risk of bleeding, with no difference in efficacy. These findings supported European dosing recommendations of 2.5mg twice daily, which differ from the U.S. recommendation of 5mg twice daily in patients with atrial fibrillation and severe chronic kidney disease.

Additionally, two recent meta-analyses included the three randomised controlled trials comparing the safety of NOACs versus warfarin. These analyses encompassed a total of 341 patients with atrial fibrillation and end-stage renal disease, with 176 in the NOAC group and 165 in the warfarin group. The results indicated that safety and efficacy outcomes were comparable, with no significant differences in stroke, mortality, or bleeding incidences.

In terms of cardiology recommendations, two meta-analyses involving a total of 10,445 patients with end-stage renal disease (ESRD) and 24,335 patients on dialysis, comparing those who received VKA with those who received no anticoagulation, revealed no significant benefit in preventing ischemic stroke but did indicate an increased risk of bleeding. Consequently, the ESC guidelines do not provide any recommendations regarding the use of NOACs in patients with atrial fibrillation (AF) who also have ESRD or are undergoing dialysis.

The results obtained from randomised controlled trials (RCTs) conducted on hemodialysis patients cannot be extrapolated to peritoneal dialysis patients. The two patient populations are distinct, as peritoneal dialysis patients do not receive heparin-based anticoagulation, which may increase the risk of bleeding events. Additionally, peritoneal dialysis patients do not have arteriovenous fistulas that could potentially lead to bleeding.

Regarding apixaban pharmacokinetics, a preliminary PK study in 2016 by Wang suggested that hemodialysis has a moderate impact on apixaban's plasma concentration. Subsequently, Mavrakanas conducted another PK study, revealing that hemodialysis was linked to supratherapeutic levels of apixaban and recommended a dose reduction.

However, as there was a lack of data on the pharmacokinetics of apixaban in end-stage renal disease (ESRD) patients undergoing peritoneal dialysis, researchers initiated the APIDP1 study with 12 peritoneal dialysis patients. The results showed a very low peritoneal dialysis apixaban clearance, resulting in significantly higher mean AUC in patients treated with PD, 73% higher (p=0.01) than the mean AUC of healthy controls matched by age, weight, and sex. Fung et al. subsequently reported similar pharmacokinetic findings : a proportion of PD patients had supratherapeutics levels even when the reduced dosage 2.5mg twice a day was use. Then Lidgard and Shen, in a 2023 editorial, emphasized the importance of reducing the apixaban dosage for stroke prevention in atrial fibrillation patients undergoing PD treatment, regardless of their age or weight.

Then, APIDP group aimed to conduct a phase III study to compare the safety of apixaban at the reduced dose to adjusted-warfarin in ESRD patients treated with chronic peritoneal dialysis. The study name is APIDP2, the protocol was prepared in accordance to Recommendations for Interventional Trials (SPIRIT) guidelines. The complete study protocol and the SPIRIT checklist are attached as supplement. The flow diagram of the study is illustrated in figure 1.

Objectives To determine in ESRD patients treated with chronic peritoneal dialysis whether apixaban 2.5mg twice daily or dose-adjusted to INR target [2-3] warfarin is safer at one year.

Methods

Trial design APIDP2 is a phase III study with a parallel enrolment, PROBE (prospective randomised open blinded-endpoint) design, one year of follow-up. Open-label administration of anticoagulation was choice because the need to adjust warfarin to targeted international normalized ratio (INR).

Setting Recruitment is scheduled to commence in June 2024 with a total of 178 randomised patients to be included. Considering the suitability of the 20 centers, it is anticipated that data collection will be completed around June 2027.

ELIGIBILITY:
Inclusion criteria

* Males and females, age at least 18 years, in ESRD treated with peritoneal dialysis for ≥ 3 months
* Patients with a history of non valvular AF treated by oral anticoagulation or patients initiating oral anticoagulation for a diagnosis of non valvular AF
* CHA2DS2-VASc score of ≥ 2.
* For women of childbearing age who are sexually active, use of an effective method of contraception for up to 10 days after the end of treatment and a negative blood pregnancy test at enrollment.
* Signature of informed consent

Exclusion criteria

* Not considered by the treating physician(s) to be candidates for oral anticoagulation (for example, hemoglobin <8.5g/dL, history of intracranial hemorrhage, active bleeding, recent gastrointestinal bleed or retroperitoneal bleed, severe hepatic impairment, or anaphylactic reaction to apixaban)
* Moderate or severe mitral stenosis
* Patients with a history of transient ischemic attack or stroke in the 3 months prior to inclusion
* Patient treated with haemodyalisis
* Conditions other than non valvular AF that require anticoagulation such as mechanical prosthetic valve, deep venous thrombosis, or pulmonary embolism
* Life expectancy < 3 months
* Anticipated kidney transplant within the next 3 months
* Individuals covered by Articles L1121-5 to L1121-8 of the French Public Health Code (corresponding to all protected persons: pregnant women, postpartum women, breastfeeding mothers, individuals deprived of their liberty by judicial or administrative decision, minors, individuals under legal protection such as guardianship or trusteeship).
* Women of childbearing age not using a highly effective contraceptive method during the study and up to 10 days after the end of treatment.
* Use of potent inducers of CYP3A4 (particularly rifampicin, phenytoin, carbamazepine, phenobarbital, or St. John's wort (Hypericum perforatum)).
* Use of CYP3A4 and P-gp inhibitors, particularly azole antifungals (ketoconazole, itraconazole, voriconazole, posaconazole, fluconazole), HIV protease inhibitors, clarithromycin, and erythromycin.
* Contraindication to anticoagulant treatment, such as antiphospholipid syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Safety primary criterion | 0-12 months
  at least one event for each participant ISTH major or clinically relevant non-major bleeding cumulated at 12 months

SECONDARY OUTCOMES:
Composite efficacy criterion | 0-12 months
  Composite criterion with at least one event :stroke or TIA, cardiovascular death, and thrombosis including myocardial infarction cumulated at 12 months

IPD SHARING:
Plan to Share IPD: Yes
Once the trial has finished and the main trial paper has been published, a fully anonymised trial data set will be available on reasonable request from Clinical Research Unit of University Hospital of Caen, Normandy, France (email: apidp2@chu-caen.fr).
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Ficheux M, Peyro-Saint-Paul L, Balayn D, Lecrux B, Brossier M, Morin A, Lanot A, Peron C, Boulanger M, Brionne M, Beygui F, Parienti JJ, Lobbedez T, Bechade C. Safety and efficacy of apixaban versus warfarin in peritoneal dialysis patients with non-valvular atrial fibrillation: protocol for a prospective, randomised, open-label, blinded endpoint trial (APIDP2). BMJ Open. 2024 Sep 20;14(9):e089353. doi: 10.1136/bmjopen-2024-089353. PMID 39306346